CLINICAL TRIAL: NCT02917369
Title: Integrative Analysis of Large-cell Lung Carcinoma
Brief Title: Integrative Analysis of Large-cell Lung Cancer
Acronym: LCLC
Status: Recruiting | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Da Fu, Principal Investigator, Shanghai 10th People's Hospital
Other Study IDs: 2016-52-Rainy
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Lung Cancer
Keywords: LCLC; Integrative Analysis; Metastasis
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Normal lung tissue: Normal lung tissue from LCLC patients
  Interventions: Other: Normal lung tissue
- LCLC tissues: LCLC tissues from LCLC patients
  Interventions: Other: Normal lung tissue
- Metastasis tissues: Metastasis tissues from LCLC patients
  Interventions: Other: Normal lung tissue

INTERVENTIONS:
Other: Normal lung tissue — The investigators will extract total protein, DNA and RNA from LCLC patients.

SUMMARY:
Integrative analysis of LCLC

DETAILED DESCRIPTION:
The investigators will analyzed proteomes of paired normal lung tissues and LCLC with or without liver metastasis, sequenced transcriptomes, perform whole exome sequencing, and single nucleotide polymorphism (SNP) array profiling for triplets, each comprising normal lung tissue, primary LCLC carcinoma, and its synchronous matched metastasis, as well as analyzed genomics of lung cancer characterized previously by The Cancer Genome Atlas (TCGA) to conduct integrated proteogenomic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 75 years with histologically proven LCLC
* No severe major organ dysfunction
* World Health Organization (WHO) performance status of 0 or 1
* No prior cancer chemotherapy

Exclusion Criteria:

* Age ≥ 76
* Severe major organ dysfunction
* WHO performance status of >1
* Prior cancer chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with large-cell lung cancer
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
5 years overall survival | 5 years

SECONDARY OUTCOMES:
5 years disease-free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Da Fu, PhD, Principal Investigator — Shanghai 10th People's Hospital
Locations (3):
- China (3):
  - Ganzhou City People's Hospital, Ganzhou, Jiangxi
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
The investigators are willing to share data.

REFERENCES:
- [Result] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787